CLINICAL TRIAL: NCT05213312
Title: A Randomized, Multicenter, Double Blind, Phase II Study of Neoadjuvant Nivolumab or Placebo Plus Chemotherapy Followed by Surgery and Adjuvant Treatment in Subjects With Resectable Esophageal Squamous Cell Carcinoma
Brief Title: Study of Neoadjuvant Nivolumab or Placebo Plus Chemotherapy Followed by Surgery and Adjuvant Treatment in Subjects With Resectable ESCC
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CA209-6KP
Record Dates: First submitted 2021-12-18; First posted 2022-01-28 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: Neoadjuvant Immunotherapy; Neoadjuvant Chemotherapy; Esophageal Squamous Cell Carcinoma; Minimally Invasive Esophagectomy
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Nivolumab; Cisplatin; Paclitaxel; Fluorouracil; Esophagectomy

STUDY DESIGN:
Intervention Model Description: Enrolled patients will receive the following medications:
  1. Neoadjuvant immunotherapy : Nivolumab, 360mg intravenous infusion (ivgtt.), on DAY1, Q3W for two cycles;
  2. Neoadjuvant chemotherapy (investigator's choice) : Cisplatin, 80 mg/m2 and Paclitaxel, 175 mg/m2 on DAY2, Q3W Or Cistaplin, 80 mg/m2 on DAY1 and 5-fluorouracil, 800 mg/m2 on DAYS1-5, Q3W for two cycles. All given intravenously.
  3. MIE : Esophagectomy plus two/three field lymphadenectomy, 4-6 weeks after neoadjuvant therapy.
  4. Adjuvant immunotherapy : 4-6 weeks after operation, (for subjects with non-pCR) Nivolumab injection, 240mg intravenous infusion, Q2W for 16 weeks, followed by 480mg intravenous infusion, Q4W. The maximum duration of adjuvant Nivolumab therapy is one year.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NIT+NCT Group (Arm A) (Experimental): 1. Neoadjuvant immunotherapy : Nivolumab, 360mg intravenous infusion (ivgtt.), on DAY1, Q3W for two cycles;
  2. Neoadjuvant chemotherapy (investigator's choice) : Cisplatin, 80 mg/m2 and Paclitaxel, 175 mg/m2 on DAY2, Q3W Or Cisplatin, 80 mg/m2 on DAY1 and 5-fluorouracil, 800 mg/m2 on DAYS1-5, Q3W for two cycles. All given intravenously.
  3. MIE : Esophagectomy plus two/three field lymphadenectomy, 4-6 weeks after neoadjuvant therapy.
  4. Adjuvant immunotherapy : 4-6 weeks after operation, (for subjects with non-pCR) Nivolumab injection, 240mg intravenous infusion, Q2W for 16 weeks, followed by 480mg intravenous infusion, Q4W. The maximum duration of adjuvant Nivolumab therapy is one year.
  Interventions: Drug: Nivolumab; Drug: Cisplatin; Drug: Paclitaxel; Drug: 5Fluorouracil; Procedure: Esophagectomy (minimally invasive)
- NCT Group (Arm B) (Placebo Comparator): 1. Placebo: NS ivgtt (dose, frequency and duration same as the Nivolumab);
  2. Neoadjuvant chemotherapy (investigator's choice) : Cisplatin, 80 mg/m2 and Paclitaxel, 175 mg/m2 on DAY2, Q3W Or Cisplatin, 80 mg/m2 on DAY1 and 5-fluorouracil, 800 mg/m2 on DAYS1-5, Q3W for two cycles. All given intravenously.
  3. MIE : Esophagectomy plus two/three field lymphadenectomy, 4-6 weeks after neoadjuvant therapy.
  4. Adjuvant immunotherapy : 4-6 weeks after operation, (for subjects with non-pCR) Nivolumab injection, 240mg intravenous infusion, Q2W for 16 weeks, followed by 480mg intravenous infusion, Q4W. The maximum duration of adjuvant Nivolumab therapy is one year.
  Interventions: Drug: Cisplatin; Drug: Paclitaxel; Drug: 5Fluorouracil; Procedure: Esophagectomy (minimally invasive)

INTERVENTIONS:
Drug: Nivolumab — Nivolumab, 360mg intravenous infusion (ivgtt.), on DAY1, Q3W for two cycles;
  Arms: NIT+NCT Group (Arm A)
Drug: Cisplatin — 80 mg/m2 on DAY2 with paclitaxel, Q3W or 80 mg/m2 on DAY1, Q3W ivgtt for two cycles
Drug: Paclitaxel — 175 mg/m2 on DAY2, with cisplatin Q3W, ivgtt for two cycles
Drug: 5Fluorouracil — 800 mg/m2 on DAYS1-5 with cisplatin, Q3W for two cycles
Procedure: Esophagectomy (minimally invasive) — 4-6 weeks after neoadjuvant therapy.

SUMMARY:
Esophageal cancer, the 7th most common cancer globally, accounts for more than half a million deaths each year. The incidence of ESCC, the most common histologic type, has been stable, whereas the incidences of esophageal and gastroesophageal junction adenocarcinomas continue to increase in Western countries.

Neoadjuvant chemoradiotherapy followed by surgery has become a standard of care for patients with locally advanced resectable esophageal or junctional cancer, especially in western countries. In Asia, nCT is considered as the standard of care for Stage II/III ESCC based on JCOG9204 and JCOG9907 trials. The superiority of nCRT/nCT, in terms of long-term survival, remains to be elucidated. For Stage II/III ESCC patients with multiple stations of lymph nodes involvement, nCT might be more appropriate for the inaccessibility of radiotherapy.

There are only limited studies on preoperative immune checkpoint inhibitor in combination with chemotherapy followed by surgery for the locally advanced ESCC. Therefore, this study intends to use Nivolumab 360 mg Q3W combined with standard chemotherapy as the neoadjuvant therapy regimen.

DETAILED DESCRIPTION:
1. Background Esophageal cancer, the 7th most common cancer globally, accounts for more than half a million deaths each year. The incidence of ESCC, the most common histologic type, has been stable, whereas the incidences of esophageal and gastroesophageal junction adenocarcinomas continue to increase in Western countries.

   Neoadjuvant chemoradiotherapy followed by surgery has become a standard of care for patients with locally advanced resectable esophageal or junctional cancer, especially in western countries. In Asia (especially Japan), nCT is considered as the standard of care for Stage II/III ESCC based on JCOG9204 and JCOG9907 trials. The superiority of nCRT/nCT, in terms of long-term survival, remains to be elucidated. For Stage II/III ESCC patients with multiple stations of lymph nodes involvement, nCT might be more appropriate for the inaccessibility of radiotherapy.

   There are only limited studies on preoperative immune checkpoint inhibitor in combination with chemotherapy followed by surgery for the locally advanced ESCC. Therefore, this study intends to use Nivolumab 360 mg Q3W combined with standard chemotherapy as the neoadjuvant therapy regimen.
2. Sample Size The planned sample size is approximately 81 subjects. The sample size calculations are based on the results of neoadjuvant therapy clinical research in our center (Department of Thoracic Surgery, Zhongshan Hospital Affiliated to Fudan University).

   In the past two years, about 85% of patients can undergo surgery and complete the entire treatment plan, combining with the results of neoadjuvant immunotherapy in lung cancer. As calculated based on an asymptotic method, 81 patients will be 2:1 randomized to Nivolumab/Chemo and Chemo group, with 80% power to detect a 21% difference in the proportion of patients achieving a pCR at a one-sided α of 0.05, assuming a pCR rate of 25% in the Nivolumab/Chemo group and 4% in the Chemo group. Considering a 10% drop rate, 90 patients will be enrolled.

   10-20 more subjects may be added to each group after the evaluation of feasibility and safety as the justification.
3. Research Process 3.1 Screening period 1) Tumor evaluation, including CT/MRI, PET/CT, endoscopy and pathological evaluation should be performed within 14 days before enrollment.

2) The following assessments should be performed within 14 days before enrollment: demographic data, concomitant diseases/treatment, full physical examination (including vital signs, KPS score, height, weight, and physical examination of the nervous system ), laboratory tests (blood routine / biochemical, fecal routine + occult blood, urine routine, coagulation function, tumor markers, thyroid function, hepatitis B and C markers, myocardial enzyme spectrum, T-SPOT, HIV antibodies), electrocardiogram (ECG), echocardiography, and pregnancy tests (for all women with menopause less than 12 months).

3) Pulmonary function tests will be performed on patients suspected or known to have severe respiratory disease or have significant respiratory symptoms unrelated to underlying cancer, including but not limited to spirometry tests and assessment of lung dispersion during the screening period to help determine if it is appropriate to participate in this study.

4) After the completion of all screening items, the researcher must review the results/data, and the subjects can only be enrolled after passing the review.

5) Subjects are required to obtain written informed consent to participate in any specific research steps. (See table below) 3.2 Treatment period Baseline assessment

1. The baseline check is performed within 7 days after signing the informed consent, and treatment must be performed within 7 days after enrollment.
2. Make the following assessments within 1 week before treatment: vital signs (temperature, blood pressure, heart rate), physical examination (including PS score, height, weight, physical examination of each system), blood routine / biochemical examination (including creatinine clearance Calculation), coagulation function, fecal routine and occult blood, urine routine and pregnancy test, tumor markers, thyroid function, hepatitis B and C markers, myocardial enzyme spectrum, T-SPOT, HIV antibodies, ECG, cardiac ultrasound, lung function.
3. When performing routine blood / biochemical examination, take 10ml blood samples for ctDNA, TCR-Seq and other analysis, and if necessary, take tissue samples for further experiments.
4. According to the above schedule, if there are already laboratory tests in the screening period, the auxiliary tests can be used as a baseline within 7 days before the start of neoadjuvant therapy, and there is no need to repeat the tests.
5. Take the chest CT, PET/CT and endoscopy as the baseline for tumor evaluation during the screening period.

After completing all screening activities and baseline assessments, eligible patients identified by the sponsor will be treated with medications, and treatment options will not be allowed to change during the study. After the investigator's first evaluation of disease progression based on RECIST, treatment can be continued if there is evidence of "pseudoprogression" and the consent of the sponsor and the patient's signing of the consent form again.

Safety will be assessed throughout the study by monitoring AE / SAE (toxicity grades are assigned according to the National Cancer Institute's Common Criteria for Adverse Events Terminology [NCI-CTCAE] version 5.0) and laboratory results. Vital signs, physical examination, changes in ECOG score, ECG results, and other tests will also be used for safety assessment.

3.3 Follow-up period after study treatment

1. Follow up at the prescribed time (recommended physical examination, tumor markers, chest CT and PET/CT). If the patient has signs of recurrence (such as related clinical manifestations), additional tumor evaluations are performed during the treatment; possible reoperations and/or further cancer treatments are also documented.
2. During the follow-up period without tumor recurrence, other cytotoxic agents are not allowed.
3. Inspection can be performed within ± 4 weeks of the specified date.
4. Patient recurrence and survival will be followed up to the patient's death, the last date on which the patient is known to survive, or 1 year after the primary effectiveness analysis.

4.Adverse Effect 4.1SERIOUS ADVERSE EVENT COLLECTION AND REPORTING All Serious Adverse Events (SAEs) that occur following the subject's written consent to participate in the study through 100 days of discontinuation of dosing must be reported to BMS Worldwide Safety, whether related or not related to study drug. If applicable, SAEs must be collected that relate to any follow-up protocol-specified procedure (eg, a follow-up skin biopsy).

4.2 NON-SERIOUS ADVERSE EVENT COLLECTION AND REPORTING The collection of non-serious AE information should begin following the subject's written consent to participate in the study. All non serious adverse events (not only those deemed to be treatment-related) should be collected continuously during the treatment period and for a minimum of 100 days following the last dose of study treatment.

Non-serious AEs should be followed to resolution or stabilization, or reported as SAEs if they become serious. Follow-up is also required for non-serious AEs that cause interruption or discontinuation of study drug and for those present at the end of study treatment as appropriate.

Non-serious Adverse Events (AE) are to be provided to BMS in aggregate via interim or final study reports as specified in the agreement or, if a regulatory requirement [eg, IND US trial] as part of an annual reporting requirement.

4.3 LABORATORY TEST ABNORMALITIES All laboratory test results captured as part of the study should be recorded following institutional procedures. Test results that constitute SAEs should be documented and reported to BMS as such.

The following laboratory abnormalities should be documented and reported appropriately:

any laboratory test result that is clinically significant or meets the definition of an SAE any laboratory abnormality that required the participant to have study drug discontinued or interrupted any laboratory abnormality that required the subject to receive specific corrective therapy.

4.4 OTHER SAFETY CONSIDERATIONS Any significant worsening noted during interim or final physical examinations, electrocardiograms, X-rays, and any other potential safety assessments, whether or not these procedures are required by the protocol, should also be recorded as a non-serious or serious AE, as appropriate, and reported accordingly.

5. Statistical analysis of research data 5.1 Statistical software All statistical analysis will be calculated using SPSS 24.0 statistical analysis software programming.

5.2 Descriptive statistics Continuous data: number of cases (number of missing cases), mean, median, standard deviation, P25, P75, minimum and maximum; Categorical data: frequency and the corresponding percentages. For primary safety endpoint, calculate the 95% CI in addition to the percentage.

5.3 Statistic inference All statistical tests are two-sided. P values less than 0.05 will be considered statistically significant. The confidence interval (CI) is 95%.

Statistical analysis for primary endpoint: pCR rates will be calculated as the proportions of the subjects in the analysis population who have a complete response in postoperative pathology.

Statistical analysis for baseline variables and secondary endpoints: the 3-year OS rates in the two treatment arms will be calculated by the Kaplan-Meier method and compared by the log rank test. The Cox proportional hazard model will be used to evaluate the survival-independent factors. Continuous variables were examined by independent sample t-test or Wilcoxon rank-sum test, and categorical variables were compared by Pearson chi-square test, Fisher's exact test or CMH chi-square test as appropriate.

5.4 Analysis of withdraw patients The number of patients who are enrolled, withdrawn, removed, completed, and number of every analysis set will be listed.

6. Research-Related Ethics 6.1 Local regulations / Helsinki Declaration Researchers should ensure that the implementation of this research is in full compliance with the principles of the Helsinki Declaration or the law of the country in the country, regardless of the country's provisions on the protection of human rights. The research must strictly follow the "ICH guideline for Good Clinical Practice" ICH Tripartite Guideline (January 1997), or local law, whichever is more stringent.

6.2 Review by Ethics Committee This protocol, written informed consent, and data directly related to the subject must be submitted to the ethics committee, and formal research can only be conducted after obtaining written approval from the ethics committee. The researcher must submit an annual research report to the Ethics Committee at least annually (if applicable). When the study is suspended and / or completed, the researcher must notify the ethics committee in writing; the researcher must promptly report all changes to the ethics committee (such as amendments to the protocol and / or informed consent) to the ethics committee, and These changes shall not be implemented until approved by the Commission, except for changes made to eliminate obvious and immediate risks to the subject. In such cases, the Ethics Committee will be notified.

6.3 Informed consent The investigator must provide the subject or his or her legal representative with an easy-to-understand, informed consent form approved by the ethics committee, and give the subject or his or her legal representative sufficient time to consider the study. Subjects shall not be enrolled until a signed written informed consent is obtained. During the participant's participation, the subject will be provided with all updated versions of informed consent and written information. The informed consent form should be kept as an important document of the clinical trial for future reference.

7. Drug and specimen management 7.1 Management of trial drugs 7.1.1 Storage Nivolumab injection is clear to opalescent, colorless to pale yellow liquid, and there may be small (rare) particles. Divided into 40mg / 4mL and 100mg / 10mL two specifications. Store and transport at 2 to 8℃ protected from light, do not freeze.

7.1.2 Inventory Nivolumab will be provided by the sponsor. The research center will confirm the receipt of nivolumab through interactive feedback technology (IRT), and confirm the transportation conditions and contents. Any medicines that are damaged or lost during transportation will be replaced. Nivolumab will be processed at the research center in accordance with the standard operating procedures of the research center or returned to the sponsor with appropriate records. The research center's method of destroying the drug must be approved by the sponsor. The research center must obtain written authorization from the sponsor before the drug is destroyed, and the drug destruction must be recorded on the appropriate form. Accurate records of all drugs received, distributed, returned, and disposed of should be recorded in the research center's drug inventory log.

7.2 Specimen management Baseline pathological specimens and blood samples of patients, surgical pathological specimens will be uniformly numbered and properly stored in the pathology laboratory of our hospital.

8. Confidentiality measures The results of research through this project may be published in medical journals, but we will keep patient information confidential as required by law, and patients 'personal information will not be leaked unless required by relevant laws. When necessary, government management departments and hospital ethics committees and their related personnel may consult patient data as required.

ELIGIBILITY:
Inclusion Criteria:

* Patients enrolled in the study must meet all of the following conditions:

  1. The patient volunteers to participate in the study, signs a consent form, has good compliance, and obeys the follow-up, and is willing and able to follow the protocol during the study.
  2. Male or female, aged ≥18 years and ≤75 years.
  3. The ECOG PS score is 0-1.
  4. Histologically-confirmed squamous cell carcinoma of the esophagus. Tumors of the esophagus are located in the thoracic cavity.
  5. Pre-treatment stage as Stage II-III (cT2N0-1M0, cT3N0-1M0, cT1-3N2M0, AJCC/UICC 8th Edition);
  6. Expected lifetime > 1 year.
  7. Adequate cardiac function. All patients should perform ECG, and those with a cardiac history or ECG abnormality should perform echocardiography with the left ventricular ejection fraction > 50 %.
  8. Adequate respiratory function with FEV1≥1.2L, FEV1%≥50% and DLCO≥50% shown in pulmonary function tests.
  9. Adequate bone marrow function (White Blood Cells >4x10^9 /L; Neutrophil >2.0×10^9 /L; Hemoglobin > 90 g/L; platelets>100x10^9 /L). AST, ALT ≤ 3 x ULN (If liver metastases exist, AST and ALT allow ≤ 5 x ULN).
  10. Adequate liver function (Total bilirubin <1.5x Upper Level of Normal (ULN); Aspartate transaminase (AST) and Alanine transaminase (ALT) <1.5x ULN).
  11. Adequate renal function (Glomerular filtration rate (CCr) >60 ml/min; serum creatinine (SCr) ≤120 μmol/L).
  12. All acute toxic effects of previous anti-cancer treatment or surgery were all relieved by NCI-CTCAE version 5.0 ≤ 1 (except for hair loss or other toxic effects that the investigator judges to have no risk to the patient's safety).
  13. Have the ability to act autonomously, have the ability to swallow pills, and have no gastrointestinal diseases that affect oral drug absorption.
  14. Agree to provide hematology and histology samples.

Exclusion Criteria:

* Patients who meet any of the following conditions will be excluded:

Patients have previously received an anti-PD-1, PD-L1 or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways.

Related to cancer:

1. Patients with non-squamous cell carcinoma histology.
2. Patients with advanced inoperable or metastatic esophageal cancer (M1).
3. Patients without qualified Pre-treatment stage.
4. Patients with another previous or current malignant disease.

Others:

1. Any patient with a significant medical condition which is thought unlikely to tolerate the therapies. Such as cardiac disease (e.g. symptomatic coronary artery disease or myocardial infarction within last 12 months), clinically-significant lung disease, clinically-significant bone marrow, liver, renal function disorder.
2. Patients who have autoimmune diseases.
3. Pregnant or lactating women and fertile women who will not be using contraception during the trial.
4. Allergy to any drugs.
5. Patients who have received or are receiving other chemotherapy, radiotherapy or targeted therapy.
6. Patients who recently or currently taking hormones or immunosuppressive agents.
7. Immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV) active infection or known HIV seropositivity; including HBV or HCV surface antigen positive (RNA).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR) rate | Up to the date of pathological reports obtained since the date of randomization, up to 12 months
  pCR rate is defined as the proportion of the subjects in the analysis population who have a complete response in postoperative pathology. It is assessed in the resected specimen following neoadjuvant therapy using standardized work up of the resection specimen in the pathology department and standardized histological criteria for tumor regression grading. The Tumor Regression Grade (TRG) is categorized as follow: grade 1, no evidence of vital residual tumor cells (pCR); grade 2, less than 10% vital residual tumor cells; grade 3, 10 to 50%; grade 4, more than 50%.

SECONDARY OUTCOMES:
R0 resection rate | Up to the date of pathological reports obtained since the date of randomization, up to 12 months
  No vital tumor is presented at the proximal, distal, or circumferential resection margin, then it is considered to be R0 resection. If a vital tumor is shown at 1 mm or less from the proximal, distal, or circumferential resection margin, it is then considered to be microscopically positive (R1).
Events-free Survival (EFS) | Up to the date of death of any causes since the date of randomization, up to 36 months
  EFS refers to the time from enrollment to the occurrence of any event, including death, disease progression, change of chemotherapy regimen, change to chemotherapy, addition of other treatments, fatal or intolerable side effects and other events.
Overall survival (OS) | Up to the date of death of any causes since the date of randomization, up to 36 months
  OS in the intent-to-treat population, which ends with the date of death of any causes since the date of randomization assessed up to 36 months. For patients alive at study closure, the survival time will be censored at time of last known survival status.
Incidence of Treatment-Emergent Adverse Events | Up to the date of death of any causes since the date of randomization, up to 36 months
  Throughout the study, NCI-CTC AE v5.0 is used to classify and record adverse drug treatment-related adverse reactions. The toxicity profile will include severity, duration, and time of occurrence.

CONTACTS AND LOCATIONS:
Locations (1):
- 180 Fenglin Road, Shanghai, China

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Kelsen DP, Ginsberg R, Pajak TF, Sheahan DG, Gunderson L, Mortimer J, Estes N, Haller DG, Ajani J, Kocha W, Minsky BD, Roth JA. Chemotherapy followed by surgery compared with surgery alone for localized esophageal cancer. N Engl J Med. 1998 Dec 31;339(27):1979-84. doi: 10.1056/NEJM199812313392704. PMID 9869669
- [Background] van Hagen P, Hulshof MC, van Lanschot JJ, Steyerberg EW, van Berge Henegouwen MI, Wijnhoven BP, Richel DJ, Nieuwenhuijzen GA, Hospers GA, Bonenkamp JJ, Cuesta MA, Blaisse RJ, Busch OR, ten Kate FJ, Creemers GJ, Punt CJ, Plukker JT, Verheul HM, Spillenaar Bilgen EJ, van Dekken H, van der Sangen MJ, Rozema T, Biermann K, Beukema JC, Piet AH, van Rij CM, Reinders JG, Tilanus HW, van der Gaast A; CROSS Group. Preoperative chemoradiotherapy for esophageal or junctional cancer. N Engl J Med. 2012 May 31;366(22):2074-84. doi: 10.1056/NEJMoa1112088. PMID 22646630
- [Background] Tepper J, Krasna MJ, Niedzwiecki D, Hollis D, Reed CE, Goldberg R, Kiel K, Willett C, Sugarbaker D, Mayer R. Phase III trial of trimodality therapy with cisplatin, fluorouracil, radiotherapy, and surgery compared with surgery alone for esophageal cancer: CALGB 9781. J Clin Oncol. 2008 Mar 1;26(7):1086-92. doi: 10.1200/JCO.2007.12.9593. PMID 18309943
- [Background] Lerut T. Neoadjuvant chemoradiotherapy followed by surgery versus surgery alone for locally advanced squamous cell carcinoma of the esophagus: the (NEOCRTEC5010) trial-a timely and welcome clinical trial from the Far East. J Thorac Dis. 2018 Nov;10(Suppl 33):S4162-S4164. doi: 10.21037/jtd.2018.10.39. No abstract available. PMID 30631582
- [Background] Turgeman I, Ben-Aharon I. Evolving treatment paradigms in esophageal cancer. Ann Transl Med. 2021 May;9(10):903. doi: 10.21037/atm.2020.03.110. PMID 34164537
- [Background] Allum WH, Stenning SP, Bancewicz J, Clark PI, Langley RE. Long-term results of a randomized trial of surgery with or without preoperative chemotherapy in esophageal cancer. J Clin Oncol. 2009 Oct 20;27(30):5062-7. doi: 10.1200/JCO.2009.22.2083. Epub 2009 Sep 21. PMID 19770374
- [Background] Ando N, Kato H, Igaki H, Shinoda M, Ozawa S, Shimizu H, Nakamura T, Yabusaki H, Aoyama N, Kurita A, Ikeda K, Kanda T, Tsujinaka T, Nakamura K, Fukuda H. A randomized trial comparing postoperative adjuvant chemotherapy with cisplatin and 5-fluorouracil versus preoperative chemotherapy for localized advanced squamous cell carcinoma of the thoracic esophagus (JCOG9907). Ann Surg Oncol. 2012 Jan;19(1):68-74. doi: 10.1245/s10434-011-2049-9. Epub 2011 Aug 31. PMID 21879261
- [Background] Sjoquist KM, Burmeister BH, Smithers BM, Zalcberg JR, Simes RJ, Barbour A, Gebski V; Australasian Gastro-Intestinal Trials Group. Survival after neoadjuvant chemotherapy or chemoradiotherapy for resectable oesophageal carcinoma: an updated meta-analysis. Lancet Oncol. 2011 Jul;12(7):681-92. doi: 10.1016/S1470-2045(11)70142-5. Epub 2011 Jun 16. PMID 21684205
- [Background] Burmeister BH, Thomas JM, Burmeister EA, Walpole ET, Harvey JA, Thomson DB, Barbour AP, Gotley DC, Smithers BM. Is concurrent radiation therapy required in patients receiving preoperative chemotherapy for adenocarcinoma of the oesophagus? A randomised phase II trial. Eur J Cancer. 2011 Feb;47(3):354-60. doi: 10.1016/j.ejca.2010.09.009. PMID 21084184
- [Background] Stahl M, Walz MK, Riera-Knorrenschild J, Stuschke M, Sandermann A, Bitzer M, Wilke H, Budach W. Preoperative chemotherapy versus chemoradiotherapy in locally advanced adenocarcinomas of the oesophagogastric junction (POET): Long-term results of a controlled randomised trial. Eur J Cancer. 2017 Aug;81:183-190. doi: 10.1016/j.ejca.2017.04.027. PMID 28628843
- [Background] von Dobeln GA, Klevebro F, Jacobsen AB, Johannessen HO, Nielsen NH, Johnsen G, Hatlevoll I, Glenjen NI, Friesland S, Lundell L, Yu J, Nilsson M. Neoadjuvant chemotherapy versus neoadjuvant chemoradiotherapy for cancer of the esophagus or gastroesophageal junction: long-term results of a randomized clinical trial. Dis Esophagus. 2019 Feb 1;32(2). doi: 10.1093/dote/doy078. PMID 30137281
- [Background] Wang H, Tang H, Fang Y, Tan L, Yin J, Shen Y, Zeng Z, Zhu J, Hou Y, Du M, Jiao J, Jiang H, Gong L, Li Z, Liu J, Xie D, Li W, Lian C, Zhao Q, Chen C, Zheng B, Liao Y, Li K, Li H, Wu H, Dai L, Chen KN. Morbidity and Mortality of Patients Who Underwent Minimally Invasive Esophagectomy After Neoadjuvant Chemoradiotherapy vs Neoadjuvant Chemotherapy for Locally Advanced Esophageal Squamous Cell Carcinoma: A Randomized Clinical Trial. JAMA Surg. 2021 May 1;156(5):444-451. doi: 10.1001/jamasurg.2021.0133. PMID 33729467
- [Background] Brahmer JR, Tykodi SS, Chow LQ, Hwu WJ, Topalian SL, Hwu P, Drake CG, Camacho LH, Kauh J, Odunsi K, Pitot HC, Hamid O, Bhatia S, Martins R, Eaton K, Chen S, Salay TM, Alaparthy S, Grosso JF, Korman AJ, Parker SM, Agrawal S, Goldberg SM, Pardoll DM, Gupta A, Wigginton JM. Safety and activity of anti-PD-L1 antibody in patients with advanced cancer. N Engl J Med. 2012 Jun 28;366(26):2455-65. doi: 10.1056/NEJMoa1200694. Epub 2012 Jun 2. PMID 22658128
- [Background] Fuchs CS, Doi T, Jang RW, Muro K, Satoh T, Machado M, Sun W, Jalal SI, Shah MA, Metges JP, Garrido M, Golan T, Mandala M, Wainberg ZA, Catenacci DV, Ohtsu A, Shitara K, Geva R, Bleeker J, Ko AH, Ku G, Philip P, Enzinger PC, Bang YJ, Levitan D, Wang J, Rosales M, Dalal RP, Yoon HH. Safety and Efficacy of Pembrolizumab Monotherapy in Patients With Previously Treated Advanced Gastric and Gastroesophageal Junction Cancer: Phase 2 Clinical KEYNOTE-059 Trial. JAMA Oncol. 2018 May 10;4(5):e180013. doi: 10.1001/jamaoncol.2018.0013. Epub 2018 May 10. PMID 29543932
- [Background] Doi T, Piha-Paul SA, Jalal SI, Saraf S, Lunceford J, Koshiji M, Bennouna J. Safety and Antitumor Activity of the Anti-Programmed Death-1 Antibody Pembrolizumab in Patients With Advanced Esophageal Carcinoma. J Clin Oncol. 2018 Jan 1;36(1):61-67. doi: 10.1200/JCO.2017.74.9846. Epub 2017 Nov 8. PMID 29116900
- [Background] Shah MA, Kojima T, Hochhauser D, Enzinger P, Raimbourg J, Hollebecque A, Lordick F, Kim SB, Tajika M, Kim HT, Lockhart AC, Arkenau HT, El-Hajbi F, Gupta M, Pfeiffer P, Liu Q, Lunceford J, Kang SP, Bhagia P, Kato K. Efficacy and Safety of Pembrolizumab for Heavily Pretreated Patients With Advanced, Metastatic Adenocarcinoma or Squamous Cell Carcinoma of the Esophagus: The Phase 2 KEYNOTE-180 Study. JAMA Oncol. 2019 Apr 1;5(4):546-550. doi: 10.1001/jamaoncol.2018.5441. PMID 30570649
- [Background] Kato K, Cho BC, Takahashi M, Okada M, Lin CY, Chin K, Kadowaki S, Ahn MJ, Hamamoto Y, Doki Y, Yen CC, Kubota Y, Kim SB, Hsu CH, Holtved E, Xynos I, Kodani M, Kitagawa Y. Nivolumab versus chemotherapy in patients with advanced oesophageal squamous cell carcinoma refractory or intolerant to previous chemotherapy (ATTRACTION-3): a multicentre, randomised, open-label, phase 3 trial. Lancet Oncol. 2019 Nov;20(11):1506-1517. doi: 10.1016/S1470-2045(19)30626-6. Epub 2019 Sep 30. PMID 31582355
- [Background] Kojima T, Shah MA, Muro K, Francois E, Adenis A, Hsu CH, Doi T, Moriwaki T, Kim SB, Lee SH, Bennouna J, Kato K, Shen L, Enzinger P, Qin SK, Ferreira P, Chen J, Girotto G, de la Fouchardiere C, Senellart H, Al-Rajabi R, Lordick F, Wang R, Suryawanshi S, Bhagia P, Kang SP, Metges JP; KEYNOTE-181 Investigators. Randomized Phase III KEYNOTE-181 Study of Pembrolizumab Versus Chemotherapy in Advanced Esophageal Cancer. J Clin Oncol. 2020 Dec 10;38(35):4138-4148. doi: 10.1200/JCO.20.01888. Epub 2020 Oct 7. PMID 33026938
- [Background] Shitara K, Ozguroglu M, Bang YJ, Di Bartolomeo M, Mandala M, Ryu MH, Fornaro L, Olesinski T, Caglevic C, Chung HC, Muro K, Goekkurt E, Mansoor W, McDermott RS, Shacham-Shmueli E, Chen X, Mayo C, Kang SP, Ohtsu A, Fuchs CS; KEYNOTE-061 investigators. Pembrolizumab versus paclitaxel for previously treated, advanced gastric or gastro-oesophageal junction cancer (KEYNOTE-061): a randomised, open-label, controlled, phase 3 trial. Lancet. 2018 Jul 14;392(10142):123-133. doi: 10.1016/S0140-6736(18)31257-1. Epub 2018 Jun 4. PMID 29880231
- [Background] Bang YJ, Ruiz EY, Van Cutsem E, Lee KW, Wyrwicz L, Schenker M, Alsina M, Ryu MH, Chung HC, Evesque L, Al-Batran SE, Park SH, Lichinitser M, Boku N, Moehler MH, Hong J, Xiong H, Hallwachs R, Conti I, Taieb J. Phase III, randomised trial of avelumab versus physician's choice of chemotherapy as third-line treatment of patients with advanced gastric or gastro-oesophageal junction cancer: primary analysis of JAVELIN Gastric 300. Ann Oncol. 2018 Oct 1;29(10):2052-2060. doi: 10.1093/annonc/mdy264. PMID 30052729
- [Background] Kang YK, Boku N, Satoh T, Ryu MH, Chao Y, Kato K, Chung HC, Chen JS, Muro K, Kang WK, Yeh KH, Yoshikawa T, Oh SC, Bai LY, Tamura T, Lee KW, Hamamoto Y, Kim JG, Chin K, Oh DY, Minashi K, Cho JY, Tsuda M, Chen LT. Nivolumab in patients with advanced gastric or gastro-oesophageal junction cancer refractory to, or intolerant of, at least two previous chemotherapy regimens (ONO-4538-12, ATTRACTION-2): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet. 2017 Dec 2;390(10111):2461-2471. doi: 10.1016/S0140-6736(17)31827-5. Epub 2017 Oct 6. PMID 28993052
- [Background] Janjigian YY, Shitara K, Moehler M, Garrido M, Salman P, Shen L, Wyrwicz L, Yamaguchi K, Skoczylas T, Campos Bragagnoli A, Liu T, Schenker M, Yanez P, Tehfe M, Kowalyszyn R, Karamouzis MV, Bruges R, Zander T, Pazo-Cid R, Hitre E, Feeney K, Cleary JM, Poulart V, Cullen D, Lei M, Xiao H, Kondo K, Li M, Ajani JA. First-line nivolumab plus chemotherapy versus chemotherapy alone for advanced gastric, gastro-oesophageal junction, and oesophageal adenocarcinoma (CheckMate 649): a randomised, open-label, phase 3 trial. Lancet. 2021 Jul 3;398(10294):27-40. doi: 10.1016/S0140-6736(21)00797-2. Epub 2021 Jun 5. PMID 34102137
- [Background] Sun JM, Shen L, Shah MA, Enzinger P, Adenis A, Doi T, Kojima T, Metges JP, Li Z, Kim SB, Cho BC, Mansoor W, Li SH, Sunpaweravong P, Maqueda MA, Goekkurt E, Hara H, Antunes L, Fountzilas C, Tsuji A, Oliden VC, Liu Q, Shah S, Bhagia P, Kato K; KEYNOTE-590 Investigators. Pembrolizumab plus chemotherapy versus chemotherapy alone for first-line treatment of advanced oesophageal cancer (KEYNOTE-590): a randomised, placebo-controlled, phase 3 study. Lancet. 2021 Aug 28;398(10302):759-771. doi: 10.1016/S0140-6736(21)01234-4. PMID 34454674
- [Background] Shitara K, Van Cutsem E, Bang YJ, Fuchs C, Wyrwicz L, Lee KW, Kudaba I, Garrido M, Chung HC, Lee J, Castro HR, Mansoor W, Braghiroli MI, Karaseva N, Caglevic C, Villanueva L, Goekkurt E, Satake H, Enzinger P, Alsina M, Benson A, Chao J, Ko AH, Wainberg ZA, Kher U, Shah S, Kang SP, Tabernero J. Efficacy and Safety of Pembrolizumab or Pembrolizumab Plus Chemotherapy vs Chemotherapy Alone for Patients With First-line, Advanced Gastric Cancer: The KEYNOTE-062 Phase 3 Randomized Clinical Trial. JAMA Oncol. 2020 Oct 1;6(10):1571-1580. doi: 10.1001/jamaoncol.2020.3370. PMID 32880601
- [Background] Kawazoe A, Yamaguchi K, Yasui H, Negoro Y, Azuma M, Amagai K, Hara H, Baba H, Tsuda M, Hosaka H, Kawakami H, Oshima T, Omuro Y, Machida N, Esaki T, Yoshida K, Nishina T, Komatsu Y, Han SR, Shiratori S, Shitara K. Safety and efficacy of pembrolizumab in combination with S-1 plus oxaliplatin as a first-line treatment in patients with advanced gastric/gastroesophageal junction cancer: Cohort 1 data from the KEYNOTE-659 phase IIb study. Eur J Cancer. 2020 Apr;129:97-106. doi: 10.1016/j.ejca.2020.02.002. Epub 2020 Mar 4. PMID 32145474
- [Background] Luo H, Lu J, Bai Y, Mao T, Wang J, Fan Q, Zhang Y, Zhao K, Chen Z, Gao S, Li J, Fu Z, Gu K, Liu Z, Wu L, Zhang X, Feng J, Niu Z, Ba Y, Zhang H, Liu Y, Zhang L, Min X, Huang J, Cheng Y, Wang D, Shen Y, Yang Q, Zou J, Xu RH; ESCORT-1st Investigators. Effect of Camrelizumab vs Placebo Added to Chemotherapy on Survival and Progression-Free Survival in Patients With Advanced or Metastatic Esophageal Squamous Cell Carcinoma: The ESCORT-1st Randomized Clinical Trial. JAMA. 2021 Sep 14;326(10):916-925. doi: 10.1001/jama.2021.12836. PMID 34519801
- [Background] Antonia SJ, Ozguroglu M. Durvalumab in Stage III Non-Small-Cell Lung Cancer. N Engl J Med. 2018 Mar 1;378(9):869-870. doi: 10.1056/NEJMc1716426. No abstract available. PMID 29490170
- [Background] Schmid P, Cortes J, Pusztai L, McArthur H, Kummel S, Bergh J, Denkert C, Park YH, Hui R, Harbeck N, Takahashi M, Foukakis T, Fasching PA, Cardoso F, Untch M, Jia L, Karantza V, Zhao J, Aktan G, Dent R, O'Shaughnessy J; KEYNOTE-522 Investigators. Pembrolizumab for Early Triple-Negative Breast Cancer. N Engl J Med. 2020 Feb 27;382(9):810-821. doi: 10.1056/NEJMoa1910549. PMID 32101663
- [Background] van den Ende T, de Clercq NC, van Berge Henegouwen MI, Gisbertz SS, Geijsen ED, Verhoeven RHA, Meijer SL, Schokker S, Dings MPG, Bergman JJGHM, Haj Mohammad N, Ruurda JP, van Hillegersberg R, Mook S, Nieuwdorp M, de Gruijl TD, Soeratram TTD, Ylstra B, van Grieken NCT, Bijlsma MF, Hulshof MCCM, van Laarhoven HWM. Neoadjuvant Chemoradiotherapy Combined with Atezolizumab for Resectable Esophageal Adenocarcinoma: A Single-arm Phase II Feasibility Trial (PERFECT). Clin Cancer Res. 2021 Jun 15;27(12):3351-3359. doi: 10.1158/1078-0432.CCR-20-4443. Epub 2021 Jan 27. PMID 33504550
- [Background] Li C, Zhao S, Zheng Y, Han Y, Chen X, Cheng Z, Wu Y, Feng X, Qi W, Chen K, Xiang J, Li J, Lerut T, Li H. Preoperative pembrolizumab combined with chemoradiotherapy for oesophageal squamous cell carcinoma (PALACE-1). Eur J Cancer. 2021 Feb;144:232-241. doi: 10.1016/j.ejca.2020.11.039. Epub 2020 Dec 26. PMID 33373868
- [Background] Ando N, Iizuka T, Ide H, Ishida K, Shinoda M, Nishimaki T, Takiyama W, Watanabe H, Isono K, Aoyama N, Makuuchi H, Tanaka O, Yamana H, Ikeuchi S, Kabuto T, Nagai K, Shimada Y, Kinjo Y, Fukuda H; Japan Clinical Oncology Group. Surgery plus chemotherapy compared with surgery alone for localized squamous cell carcinoma of the thoracic esophagus: a Japan Clinical Oncology Group Study--JCOG9204. J Clin Oncol. 2003 Dec 15;21(24):4592-6. doi: 10.1200/JCO.2003.12.095. PMID 14673047
- [Background] Urba SG, Orringer MB, Turrisi A, Iannettoni M, Forastiere A, Strawderman M. Randomized trial of preoperative chemoradiation versus surgery alone in patients with locoregional esophageal carcinoma. J Clin Oncol. 2001 Jan 15;19(2):305-13. doi: 10.1200/JCO.2001.19.2.305. PMID 11208820
- [Background] Burmeister BH, Smithers BM, Gebski V, Fitzgerald L, Simes RJ, Devitt P, Ackland S, Gotley DC, Joseph D, Millar J, North J, Walpole ET, Denham JW; Trans-Tasman Radiation Oncology Group; Australasian Gastro-Intestinal Trials Group. Surgery alone versus chemoradiotherapy followed by surgery for resectable cancer of the oesophagus: a randomised controlled phase III trial. Lancet Oncol. 2005 Sep;6(9):659-68. doi: 10.1016/S1470-2045(05)70288-6. PMID 16129366
- [Background] Lordick F, Mariette C, Haustermans K, Obermannova R, Arnold D; ESMO Guidelines Committee. Oesophageal cancer: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2016 Sep;27(suppl 5):v50-v57. doi: 10.1093/annonc/mdw329. No abstract available. PMID 27664261
- [Background] Smyth EC, Gambardella V, Cervantes A, Fleitas T. Checkpoint inhibitors for gastroesophageal cancers: dissecting heterogeneity to better understand their role in first-line and adjuvant therapy. Ann Oncol. 2021 May;32(5):590-599. doi: 10.1016/j.annonc.2021.02.004. Epub 2021 Feb 17. PMID 33609722
- [Background] Zhang X, Schwartz JC, Guo X, Bhatia S, Cao E, Lorenz M, Cammer M, Chen L, Zhang ZY, Edidin MA, Nathenson SG, Almo SC. Structural and functional analysis of the costimulatory receptor programmed death-1. Immunity. 2004 Mar;20(3):337-47. doi: 10.1016/s1074-7613(04)00051-2. PMID 15030777
- [Background] Nishimura H, Honjo T. PD-1: an inhibitory immunoreceptor involved in peripheral tolerance. Trends Immunol. 2001 May;22(5):265-8. doi: 10.1016/s1471-4906(01)01888-9. PMID 11323285
- [Background] Konishi J, Yamazaki K, Azuma M, Kinoshita I, Dosaka-Akita H, Nishimura M. B7-H1 expression on non-small cell lung cancer cells and its relationship with tumor-infiltrating lymphocytes and their PD-1 expression. Clin Cancer Res. 2004 Aug 1;10(15):5094-100. doi: 10.1158/1078-0432.CCR-04-0428. PMID 15297412
- [Background] Thompson RH, Gillett MD, Cheville JC, Lohse CM, Dong H, Webster WS, Krejci KG, Lobo JR, Sengupta S, Chen L, Zincke H, Blute ML, Strome SE, Leibovich BC, Kwon ED. Costimulatory B7-H1 in renal cell carcinoma patients: Indicator of tumor aggressiveness and potential therapeutic target. Proc Natl Acad Sci U S A. 2004 Dec 7;101(49):17174-9. doi: 10.1073/pnas.0406351101. Epub 2004 Nov 29. PMID 15569934
- [Background] Ohigashi Y, Sho M, Yamada Y, Tsurui Y, Hamada K, Ikeda N, Mizuno T, Yoriki R, Kashizuka H, Yane K, Tsushima F, Otsuki N, Yagita H, Azuma M, Nakajima Y. Clinical significance of programmed death-1 ligand-1 and programmed death-1 ligand-2 expression in human esophageal cancer. Clin Cancer Res. 2005 Apr 15;11(8):2947-53. doi: 10.1158/1078-0432.CCR-04-1469. PMID 15837746
- [Background] Boussiotis VA. Molecular and Biochemical Aspects of the PD-1 Checkpoint Pathway. N Engl J Med. 2016 Nov 3;375(18):1767-1778. doi: 10.1056/NEJMra1514296. No abstract available. PMID 27806234
- [Background] Brahmer JR, Drake CG, Wollner I, Powderly JD, Picus J, Sharfman WH, Stankevich E, Pons A, Salay TM, McMiller TL, Gilson MM, Wang C, Selby M, Taube JM, Anders R, Chen L, Korman AJ, Pardoll DM, Lowy I, Topalian SL. Phase I study of single-agent anti-programmed death-1 (MDX-1106) in refractory solid tumors: safety, clinical activity, pharmacodynamics, and immunologic correlates. J Clin Oncol. 2010 Jul 1;28(19):3167-75. doi: 10.1200/JCO.2009.26.7609. Epub 2010 Jun 1. PMID 20516446
- [Background] Rizvi NA, Hellmann MD, Brahmer JR, Juergens RA, Borghaei H, Gettinger S, Chow LQ, Gerber DE, Laurie SA, Goldman JW, Shepherd FA, Chen AC, Shen Y, Nathan FE, Harbison CT, Antonia S. Nivolumab in Combination With Platinum-Based Doublet Chemotherapy for First-Line Treatment of Advanced Non-Small-Cell Lung Cancer. J Clin Oncol. 2016 Sep 1;34(25):2969-79. doi: 10.1200/JCO.2016.66.9861. Epub 2016 Jun 27. PMID 27354481
- [Background] Yamamoto S, Kato K, Daiko H, Kojima T, Hara H, Abe T, Tsubosa Y, Nagashima K, Aoki K, Mizoguchi Y, Kitano S, Yachida S, Shiba S, Kitagawa Y. Feasibility study of nivolumab as neoadjuvant chemotherapy for locally esophageal carcinoma: FRONTiER (JCOG1804E). Future Oncol. 2020 Jul;16(19):1351-1357. doi: 10.2217/fon-2020-0189. Epub 2020 May 12. PMID 32396014
- [Background] Dueck AC, Mendoza TR, Mitchell SA, Reeve BB, Castro KM, Rogak LJ, Atkinson TM, Bennett AV, Denicoff AM, O'Mara AM, Li Y, Clauser SB, Bryant DM, Bearden JD 3rd, Gillis TA, Harness JK, Siegel RD, Paul DB, Cleeland CS, Schrag D, Sloan JA, Abernethy AP, Bruner DW, Minasian LM, Basch E; National Cancer Institute PRO-CTCAE Study Group. Validity and Reliability of the US National Cancer Institute's Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE). JAMA Oncol. 2015 Nov;1(8):1051-9. doi: 10.1001/jamaoncol.2015.2639. PMID 26270597
- [Derived] Jiao H, Lin S, Gu J, Jiang D, Cui P, Huang Z, Fang Y, Wang H, Lin M, Tang H, Jiang T, Lin G, Zhang S, Yin H, Liang F, Wang J, Fan X, Qiu F, Yang Y, Li Z, Li B, Xiang J, Leng X, Han Y, Li C, Ai L, Hou Y, Wang G, Zhang Z, Cai S, Liu T, Yin J, Tan L. Perioperative nivolumab and chemotherapy in locally advanced squamous cell carcinoma of the oesophagus: a randomized multicentre phase 2 study with circulating tumor DNA dynamics monitoring. Mol Cancer. 2025 May 15;24(1):143. doi: 10.1186/s12943-025-02332-8. PMID 40375301
- [Derived] Al-Batran SE, Koch C. Neoadjuvant therapy for oesophageal cancer: refining the armamentarium. Lancet. 2024 Jul 6;404(10447):5-7. doi: 10.1016/S0140-6736(24)01084-5. Epub 2024 Jun 11. No abstract available. PMID 38876135
- [Derived] Yin J, Lin S, Fang Y, Jiao H, Chen Z, Tang H, Gu J, Zhang S, Sun L, Li Y, Han Y, Chen Q, Chen H, Li Z, Tan L. Neoadjuvant therapy with immunoagent (nivolumab) or placebo plus chemotherapy followed by surgery and adjuvant treatment in subjects with resectable esophageal squamous cell carcinoma: study protocol of a randomized, multicenter, double blind, phase II trial (NATION-2203 trial). J Thorac Dis. 2023 Feb 28;15(2):718-730. doi: 10.21037/jtd-22-1789. Epub 2023 Feb 8. PMID 36910109